CLINICAL TRIAL: NCT03150836
Title: Multi-Institutional Phase II Study of Radiation Therapy and Anti-PD-L1 Checkpoint Inhibition (Durvalumab) With or Without Anti-CTLA-4 Inhibition (Tremelimumab) in Patients With Unresectable, Muscle-Invasive or Metastatic Urothelial Bladder Cancer That Are Ineligible or Refusing Chemotherapy
Brief Title: Radiation Therapy and Durvalumab, With or Without Tremelimumab, in Patients With Bladder Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Co-PI Albert Chang relocating to UCLA. IND will transfer to UCLA. UCSF will not participate.
Sponsor: Terence Friedlander, MD (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor-Investigator, Terence Friedlander, MD, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16529
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; urothelial
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; tremelimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Safety Lead-In, Regimen A1 Durvalumab + RT (Experimental): Durvalumab 1500 mg will be delivered via IV infusion q4wk. Radiation Therapy (RT) will be delivered beginning on day 8 ± 3 of durvalumab. RT (33Gy delivered as 6.6Gy x 5 fractions) should be completed within 14 days from the start of RT ideally over 5 consecutive days. Durvalumab 1500 mg q4wk will be continued to complete either 13 total cycles OR until disease progression, unacceptable toxicity, or patient withdrawal from study, whichever comes first.
  Interventions: Drug: Durvalumab; Radiation: Radiation Therapy
- Safety Lead-In, Regimen A2 Durvalumab + RT (Experimental): In cohort A2 the dose of radiation will be decreased to a total dose of 30 Gy administered in 5 fractions of 6 Gy. Durvalumab 1500 mg will be delivered via IV infusion q4wk. Radiation Therapy (RT) will be delivered beginning on day 8 ± 3 of durvalumab. RT (30 Gy delivered as 6.0Gy x 5 fractions) should be completed within 14 days from the start of RT ideally over 5 consecutive days. Durvalumab 1500 mg q4wk will be continued to complete either 13 total cycles OR until disease progression, unacceptable toxicity, or patient withdrawal from study, whichever comes first.
  Interventions: Drug: Durvalumab; Radiation: Radiation Therapy
- Safety Lead-In, Regimen B1 Durvalumab + Tremelimumab + RT (Experimental): Tremelimumab 75 mg will be administered via IV infusion q4wk for 2 cycles with durvalumab 1500 mg via IV infusion. Radiation Therapy (RT), at the optimal dose determined in the safety lead-in from Regimen A, will be delivered beginning on day 8 ± 3 of durvalumab. After two doses of tremelimumab and durvalumab, durvalumab 1500 mg q4wk will be continued to complete either 13 total cycles of durvalumab OR until disease progression, unacceptable toxicity, or patient withdrawal from study, whichever comes first.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Radiation Therapy
- Safety Lead-In, Regimen B2 Durvalumab + Tremelimumab + RT (Experimental): Tremelimumab 75 mg will be administered via IV infusion q4wk for 1 cycle with durvalumab 1500 mg via IV infusion. Radiation Therapy (RT), at the optimal dose determined in the safety lead-in from Regimen A, will be delivered beginning on day 8 ± 3 of durvalumab. After one dose of tremelimumab and durvalumab, durvalumab 1500 mg q4wk will be continued to complete either 13 total cycles of durvalumab OR until disease progression, unacceptable toxicity, or patient withdrawal from study, whichever comes first.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Radiation Therapy
- Expansion Cohort, Regimen A: Durvalumab + RT (Experimental): Durvalumab 1500 mg will be delivered via IV infusion q4wk. Radiation Therapy (RT) will be delivered beginning on day 8 ± 3 of durvalumab. RT (either 33Gy delivered as 6.6Gy x 5 fractions or 30 Gy delivered as 6.0 Gy x 5 fractions, as determined during the safety lead-in for Regimen B) should be completed within 14 days from the start of RT ideally over 5 consecutive days. Durvalumab 1500 mg q4wk will be continued to complete either 13 total cycles OR until disease progression, unacceptable toxicity, or patient withdrawal from study, whichever comes first.
  Interventions: Drug: Durvalumab; Radiation: Radiation Therapy
- Expansion Cohort Regimen B: Durvalumab + Tremelimumab + RT (Experimental): Tremelimumab 75 mg will be administered via IV infusion q4wk for 1 or 2 cycles (as determined during the safety lead-in for Regimen B) with durvalumab 1500 mg via IV infusion. Radiation Therapy (RT), at the optimal dose determined in the safety lead-in from Regimen A, will be delivered beginning on day 8 ± 3 of durvalumab. After 1 or 2 doses of tremelimumab and durvalumab, durvalumab 1500 mg q4wk will be continued to complete either 13 total cycles of durvalumab OR until disease progression, unacceptable toxicity, or patient withdrawal from study, whichever comes first.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Durvalumab — All participants will receive durvalumab 1500 mg via IV infusion every 4 weeks for up to 13 doses.
  Other Names: Imfinzi
Drug: Tremelimumab — Participants receiving Regimen B (safety lead-in or expansion cohort) will be administered tremelimumab 75 mg via IV infusion every 4 weeks for 1 cycle or 2 cycles.
  Arms: Expansion Cohort Regimen B: Durvalumab + Tremelimumab + RT; Safety Lead-In, Regimen B1 Durvalumab + Tremelimumab + RT; Safety Lead-In, Regimen B2 Durvalumab + Tremelimumab + RT
Radiation: Radiation Therapy — In all arms of the study, participants will receive 5 fractions of radiation. The radiation dose will either be 6.6 Gy for a total dose of 33 Gy, or 6.0 Gy for a total dose of 30 Gy.

SUMMARY:
This is a multi-site, randomized, prospective, open-label phase II study. Patients in this study will have localized (cT3-cT4), or metastatic bladder cancer with a symptomatic, intact primary bladder tumor. In this study, patients will undergo stereotactic body radiation therapy (SBRT) to the bladder tumor and will receive durvalumab with or without tremelimumab.

DETAILED DESCRIPTION:
The study will commence with a safety lead-in phase at UCSF in which 6 patients are accrued to Regimen A1 (RT + durvalumab). If this is not tolerated then an alternative Regimen A2, containing a lower total radiation dose will accrue 6 patients. If either A1 or A2 is tolerated then patients will be accrued to Regimen B1 (durvalumab, tremelimumab x 2 doses, and RT dose determined from Regimen A) following a 3+3 design for safety. If Regimen B1 is not tolerated an alternative Regimen B2 (durvalumab, tremelimumab x 1 dose, and RT dose determined from regimen A) will accrue following a 3+3 design for safety.

After the safety lead-in for each group is completed, an expansion cohort will accrue patients. In this expansion cohort, patients will be randomized 1:1 to be treated with either regimen A or regimen B dose selected from the safety lead-in stratified by patient population (localized patients and metastatic patients).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
2. Locally advanced (cT3 or cT4) or metastatic (N+ or M+) urothelial bladder cancer. Mixed histologies with predominant urothelial pattern are allowed
3. If metastatic disease present patients must have an intact, symptomatic bladder tumor, appropriate for palliative RT to the bladder.
4. Measurable metastatic disease according to RECIST v1.1 criteria. Thus, patients with metastatic disease must have at least 1 lesion, not previously irradiated, that can be accurately measured at baseline as at least 10 mm in the longest diameter (except lymph nodes which must have a short axis greater than or equal to 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurement as per RECIST v1.1 guidelines.
5. Age greater than or equal to 18 years at time of study entry
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Life expectancy of at least 12 weeks
8. Patients with non-metastatic bladder cancer must be ineligible for cystectomy in the opinion of the treating investigator.
9. Patients must be ineligible for cisplatin-based chemotherapy. The reason for cisplatin ineligibility must be documented. Cisplatin ineligibility is defined as meeting 1 of the following criteria:

   * Creatinine clearance (calculated or measured) less than 60 mL/min
   * Common Terminology Criteria for Adverse Events (CTCAE) Grade greater than or equal to 2 audiometric hearing loss
   * CTCAE Grade 2 or higher peripheral neuropathy
   * New York Heart Association Class III heart failure
   * Any other criteria deemed by the investigator to make the patient unsuitable for cisplatin-based chemotherapy.
10. Subjects must consent to provide an archived tumor specimen from within 12 months prior to study entry (ie, from subject signing consent to participate in the study) for immunologic characterization. If not available, subjects should have at least 1 lesion amenable to biopsy and consent to provide a pre-treatment fresh biopsy. Tumor lesions used for biopsy should not be lesions used as target lesions. Additional archival tissue from beyond 12 months prior to study entry is also requested, if available, to support exploratory analyses.
11. Adequate normal organ and marrow function as defined below:

    * Hemoglobin greater than or equal to 9.0 g/dL
    * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L (greater than 1500 per mm3)
    * Platelet count greater than or equal to 100 x 109/L (greater than100,000 per mm3)
    * Serum bilirubin less than or equal to 1.5 x institutional upper limit of normal (ULN). [This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician].
    * AST (SGOT)/ALT (SGPT) less than or equal to 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be less than or equal to 5x ULN.
    * Serum creatinine CL greater than 30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance. Serum creatine measurement is the preferred measurement for determining creatinine clearance.

    Males:

    Creatinine CL (mL/min) = [Weight (kg) x (140 - Age)] / [72 x serum creatinine (mg/dL)]

    Females:

    Creatinine CL (mL/min) = 0.85 x [Weight (kg) x (140 - Age)] / [72 x serum creatinine (mg/dL)]
12. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: At least 60 years old and no menses for at least 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women less than 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women greater than or equal to 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses more than 1 year ago, had chemotherapy-induced menopause with last menses more than 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visit and examinations and follow-up.

Exclusion Criteria:

1. ECOG PS 2 or higher
2. Upper tract-only or urethral-only urothelial cancer
3. Prior cystectomy or definitive RT to the bladder.
4. Prior systemic chemotherapy for bladder cancer
5. History of autoimmune disease, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Subjects with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
   * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are not excluded.
   * Patients with controlled type 1 diabetes mellitus on a stable dose of insulin regimen are not excluded.
   * Any chronic skin condition that does not require systemic therapy are not exluded
   * Patients without active autoimmune disease in the last 5 years may be included after consultation with the study physician.
7. Patients with HIV, active hepatitis B (HBV) or active hepatitis C (HCV)

   * Patients with past HBV infection or resolved HBV infection, defined as the presence of hepatitis B core antibody (HBc Ab) and absence of hepatitis B surface antigen (HBsAg) are eligible. HBV DNA must be obtained in these patients prior to day 1 of therapy, but detection of HBV DNA in these patients will not exclude study participation.
   * Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
8. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
9. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
10. Previous IP assignment in the present study
11. Current enrollment/participation in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.
12. Prior exposure to immune-mediated therapy, including but not limited to, durvalumab, tremelimumab, other anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies, and therapeutic anticancer vaccines. Prior BCG or intravestical immune therapy (ie interferon) is not an exclusion to study participation.
13. Prior radiation therapy to the abdomen or pelvis.
14. Any concurrent systemic chemotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (i.e. hormonal replacement therapy) is acceptable.
15. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note biopsy and TURBT of the primary tumor is acceptable.
16. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease for at least 5 years before the first dose of study drug and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ. (Optional criteria that are dependent on the patient population under investigation.)
    * Patients with incidental finding of early stage prostate cancer will not be eligible.
17. QT interval corrected for heart rate using Fridericia's formula (QTcF) greater than or equal to 470 ms calculated. Any clinically significant abnormalities detected require triplicate ECG results and a mean QT interval corrected for heart rate using Fridericia's formula (QTcF) greater than or equal to 470 ms calculated from 3 ECGs).
18. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
19. History of primary immunodeficiency
20. History of allogeneic organ transplant
21. History of hypersensitivity to durvalumab, tremelimumab, or any excipient
22. History of hypersensitivity to the combination
23. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
24. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice).
25. History of leptomeningeal carcinomatosis
26. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
27. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
28. Brain metastases or spinal cord compression unless the patient's condition is stable (asymptomatic, no evidence of new or emerging brain metastases) and off steroids for at least 14 days prior to the start of study treatment. Following radiotherapy and/or surgery, patients with suspected brain metastases at screening should have an MRI (preferred)/CT, preferably with IV contrast.
29. Subjects with uncontrolled seizures.
30. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity according to NCI CTCAE v. 4.03 criteria | Over the duration of the study, which is estimated to be approximately 50 months.
  Safety profile
Progression-free survival (PFS) | Over the duration of the study, which is estimated to be approximately 50 months.
  PFS will be determined from first day of treatment to date of progression. Progression will be defined based on RECIST 1.1

SECONDARY OUTCOMES:
Local control at the primary irradiated site | Over the duration of the study, which is estimated to be approximately 50 months.
  As determined by RECIST v 1.1 from the date of randomization to the date of first local progression.
Pathologic Complete Response (CR) rate of primary irradiated tumor | Over the duration of the study, which is estimated to be approximately 50 months.
  As determined by post-treatment biopsy or TURBT in evaluable patients.
Overall response rate (ORR) | Over the duration of the study, which is estimated to be approximately 50 months.
  The ORR will be as determined by RECIST v 1.1. The ORR will be defined as the number (%) of patients with at least 1 visit response of CR or Partial Response (PR).
Abscopal response (in patients with metastatic disease) | Over the duration of the study, which is estimated to be approximately 50 months.
  As determined by RECIST v 1.1 with response (PR and CR) sites away from the primary irradiated tumor.
Duration of response | Over the duration of the study, which is estimated to be approximately 50 months.
  Defined as the time from the date of the first documented response until the first date of documented progression or death.
Disease-specific survival | Over the duration of the study, which is estimated to be approximately 50 months.
  Defined as the time from the first day of treatment to the date of death related to treatment and/or disease.
Overall survival | Over the duration of the study, which is estimated to be approximately 50 months.
  Defined as the time from the first day of treatment to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Friedlander, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No